CLINICAL TRIAL: NCT03184129
Title: Safety and Efficacy of Newly Developed Knee Prosthesis for Knee Arthroplasty: a Prospective, Single-center, Randomized, Positive Parallel Controlled, Non-inferiority Clinical Trial
Brief Title: Safety and Efficacy of Newly Developed Knee Prosthesis for Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taihe Hospital (Other)
Responsible Party: Principal Investigator, Taifang Gong, Principal Investigator, Taihe Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TaiheH_001
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Knee Disease
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): Patients with knee disease who will undergo knee arthroplasty will be randomized into trial group. The patients from the trial group will receive knee arthroplasty with knee prostheses purchased from Wuhan Yijiabao Biomaterial Co., Ltd., Wuhan, China (newly developed).
  Interventions: Device: trial group
- control group (Experimental): Patients with knee disease who will undergo knee arthroplasty will be randomized into control group. The patients from the control group will receive knee arthroplasty with knee prostheses purchased from Beijing AKEC Medical Co., Ltd., Beijing, China (approved by China Food and Drug Administration).
  Interventions: Device: control group

INTERVENTIONS:
Device: trial group — Patients with knee disease who will undergo knee arthroplasty will be randomized into trial group. The patients from the trial group will receive newly developed knee arthroplasty with knee prostheses purchased from Wuhan Yijiabao Biomaterial Co., Ltd..
  Other Names: newly developed knee prosthesis
  Arms: trial group
Device: control group — Patients with knee disease who will undergo knee arthroplasty will be randomized into control group. The patients from the control group will receive knee arthroplasty with knee prostheses purchased from Beijing AKEC Medical Co., Ltd., Beijing, China (approved by China Food and Drug Administration).
  Other Names: knee prosthesis approved by CFDA
  Arms: control group

SUMMARY:
To verify and assess the safety and efficacy of newly developed knee prosthesis (Wuhan Yijiabao Biomaterial Co., Ltd.) in total knee arthroplasty.

DETAILED DESCRIPTION:
Background Total knee arthroplasty is one of major means in the treatment of end-stage knee disease. Therefore, there is an urgent need to develop a safe, effective, high-quality and inexpensive knee prosthesis so as to meet the huge demand for replacement repair in patients with knee diseases in China.

Combined with international advanced design concept, Wuhan Yijiabao Biomaterial Co., Ltd. of China has developed a new set of knee prosthesis system with cobalt-chromium-molybdenum alloy and high cross-linked polyethylene as the main materials. This knee prosthesis system contains femoral condyle, meniscus, tibial tray, and patella. This system uses cobalt-chrome-molybdenum and high cross-linked polyethylene as the active friction interface, which has excellent wear resistance, and provides an ideal treatment for patients with knee diseases. The difference in the efficacy and safety between widely used knee prosthesis and this newly developed knee prosthesis after total knee arthroplasty deserves further verification by randomized controlled clinical trial.

Data collection, management, analysis, and open access

* Data collection: The researchers will fill out a papery case report form for each case. The case report form will be truthfully and carefully recorded in detailed to ensure that the case report form is complete, authentic and reliable.
* Data management: The entire experiment will strictly enforce quality management specification for clinical trials. All papery case report form records will be complete, true, clear and objective. All data will be input to the computer, locked and stored. The completed case report form will be reviewed by the inspector. The first page of the case report form will be handed over to the data manager for data entry and management. From then on, the contents of the case report form will not be altered.
* Data analysis: After the test plan has been determined, the statisticians will be responsible for consultation with the major researchers and formulate a statistical analysis plan. All data will be analyzed using SAS9.3 software. Statistical analysis includes actual number of participants in the two groups, the conditions of dropped-out and eliminated cases, demographic and other baseline characteristics, efficacy analysis, and safety analysis. Besides the statistical methods listed below, detailed and additional exploratory analyses may be necessary, and may be identified in the study report and analysis plan.
* Data open access: If the researchers want to publish or disclose the results obtained from the products of this clinical trial, they must have the prior written consent of the sponsor. The sponsor will review and reply the contents of the proposed disclosure within 30 working days. Without the consent of the researchers, the sponsor will not use the name of the researcher in the advertising of the test equipment. However, in the case of a clinical trial of the test instrument and the submission of a production license to the China Food and Drug Administration, the sponsor can, without the consent of the researchers, directly use all the results obtained from the clinical trial.

Quality control The researchers will strictly comply with the state regulations on the clinical trials of medical devices and the relevant operating procedures. Institutional and personnel requirements: The research center must obtain the qualification of the national clinical drug testing institution in orthopedics. Before the trial, the related personnels will be trained, including clinical protocols, informed procedures, equipment use, and file filling. During the trial, the researchers and test-related personnels will receive targeted training according to the clinical situation.

Statistical analysis

1. Data will be analyzed using SAS 9.3 software.
2. Measurement data will be expressed as means ± standard deviation and minimums and maximums. Measurement data and registration data will be described by frequency.
3. The difference in the excellent and good rate between the trial and control groups and its 95%CI will be calculated. The lower limit greater than -10.0% can be considered as non-inferiority. Measurement data will be compared using two-sample t-test or Mann Whitney U rank sum test between the two groups. Intergroup comparison will be conducted using Pearson's chi-squared test or Fisher's exact test. Ranked data in both groups will be analyzed using Wilcoxon rank-sum test or Cochran-Mantel-Haenszel test.
4. Efficacy evaluation: The excellent and good rate between the trial and control groups will receive non-inferiority trial. Non-inferiority margin δ = 10.0%. The test is assumed to be:

   H0: Difference of excellent and good rate between the trial and control groups (πT-πC) ≤ -δ H1: Difference of excellent and good rate between the trial and control groups (πT-πC) > -δ Cochran-Mantel-Haenszel test will be considered to compare the difference of excellent and good rate between the trial and control groups and to calculate the lower limit of 95%CI on one side. The lower limit greater than -10.0% will be considered as non-inferiority.
5. Safety evaluation: The incidence of adverse events between the two groups will be compared using chi-square test.
6. Data processing for patients undergoing arthroplasty on both knees: If the indicators are evaluated separately on both sides, the data on one side are included in the statistical analysis set under two conditions. When both knees are operated simultaneously, data of the knee with poor postoperative efficacy will be taken into the analysis set. When both knees are operated in different stages, data of the knee undergoing the second operation will be taken into the analysis set.
7. Report deviated from the original statistical plan: In case of "incomplete implementation of statistical analysis plan", the change procedure will be applied in advance. For example, changes in the statistical plan shall be faithfully recorded in the statistical analysis plan, including place, reason and time.
8. Subjects' selection criteria and set analysis:

Full analysis set: According to the intention-to-treat principle, the data sets consisting of subjects who participated in the treatment and had baseline efficacy evaluation. For subjects who do not have the overall efficacy evaluation, the last observation carry forward principle will be used for data conversion.

Per protocol set: Patients have finished the trial and breach of inclusion criteria or exclusion criteria.

Safety set: All subjects using the test apparatus and who have at least one baseline safety evaluation. The efficacy analysis will be carried out on the basis of full analysis set and per protocol set. All baseline demographic data analyses will be conducted on the full analysis set, and security evaluation will be carried out on the safety set.

ELIGIBILITY:
Inclusion Criteria:

* At least one knee disease: Primary or secondary knee osteoarthritis, traumatic arthritis, rheumatoid arthritis or ankylosing spondylitis and other systemic diseases involving the knee, degenerative arthritis, tumor resection of the knee, varus or valgus correction of the knee and fracture of the knee joint
* At the age of at least 35 years old, irrespective of sex
* Bone is mature; that is, knee X-ray shows epiphyseal closure
* First total knee arthroplasty
* Willing and able to sign informed consent

Exclusion Criteria:

* Neuromuscular dysfunction (such as paralysis, rhabdomyolysis, or abductor weakness) can lead to instability or gait abnormalities in the knee after surgery
* Mentally incapable or unable to understand the requirements for participation in research
* Expected to be incompatible (such as alcohol, drug addicts, drug abusers; unwilling to accept a 12-month study plan; the patient's expected value is unrealistic or the patient has a clear emotional problem)
* Allergic to one or more implants
* An active infection lesion in the knee joint or other parts of the body
* Severe osteoporosis, bone defect, metabolic bone disease and radioactive bone disease around the knee joint
* Frail or unable to tolerate surgery because of other diseases of the body, or a life expectancy of less than 2 years
* A pregnant or lactating woman or woman expecting to have children
* The combination of other diseases restricts its participation in the study; failure to follow up or influence the scientific nature and integrity of the study (for example, other lower joint (ankle) disorders cause severe functional impairment and influence assessment; other primary joints (knee and hip) have been implanted with joint prostheses)
* Participation in other clinical trials of drug, biological agents or instruments, and have not reach the research time limit

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Hospital for Special Surgery Knee Scores | at postoperative 12 months (±15 days)
  To evaluate the recovery of knee function.That is the percentage of the number of patients with excellent and good HSS scores after surgery in each group. HSS scores: total score is 100. Excellent: 85-100; good: 70-84; average: 60-69; poor: less than 59.

SECONDARY OUTCOMES:
X-ray | at postoperative 12 months (±15 days)
  To assess the morphology of the knee after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Taifang Gong, Ph.D, Principal Investigator — Taihe Hospital
Locations (1):
- Taihe Hospital, Shiyan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided